CLINICAL TRIAL: NCT06968897
Title: Neurological Development in Toddlers After Maternal SARS-CoV-2 Infection During Pregnancy - A Follow-Up to the Covid-19 Related Obstetric and Neonatal Outcome Study in Germany (CRONOS) With a Dedicated Focus on Child Health
Brief Title: Neurological Development In Toddlers After Maternal SARS-CoV-2 Infection During Pregnancy
Acronym: CRONOS-Kids
Status: Enrolling by invitation | Type: Observational
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Dr. med. Nadine Mand, Dr. med. Nadine Mand, Philipps University Marburg
Other Study IDs: AZ 114/22
Record Dates: First submitted 2025-04-16; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: SARS CoV-2; Developmental Disorder; Pregnancy Related
Keywords: SARS-CoV-2; Children; Development; pregnancy
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed intrauterine to SARS-CoV-2: Toddlers exposed to SARS-CoV-2 (VOC alpha or delta) during their mothers' pregnancy.
- Not exposed to SARS-CoV-2: Toddlers NOT exposed to SARS-CoV-2 (VOC alpha or delta) during their mothers' pregnancy.

SUMMARY:
Severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2) is a virus that causes neurological symptoms in a significant proportion of patients in addition to respiratory symptoms. Intrauterine exposure to the virus has been demonstrated to exert a detrimental effect on the developing nervous system. However, developmental disorders frequently remain undetected until late infancy or early childhood. Consequently, there is a paucity of published data on neurodevelopment in young children following SARS-CoV-2 infection of their pregnant mothers.

To this end, detailed data from children aged 36-60 months exposed to SARS-CoV-2 in utero will be compared with unexposed children of the same age on several clinical outcome parameters. Data in this cohort study will be adjusted for possible confounding variables, such as gestational age at birth, sex, or umbilical arterial pH, in order to investigate a relative risk of intrauterine SARS-CoV-2 infection on clinical outcomes, such as child development. Furthermore, the potential protective effect of SARS-CoV-2 vaccination during pregnancy will be investigated.

This study will provide significant data on the clinical outcomes of children exposed perinatally to SARS-CoV-2. The findings will enable healthcare providers to establish a risk score-adapted follow-up strategy for the general paediatric population of infants.

DETAILED DESCRIPTION:
In Utero Exposure to SARS-CoV-2 - the CRONOS registry The "COVID-19 Related Obstetric and Neonatal Outcome Study" (CRONOS) investigated the short-term effects of SARS-CoV-2 infections on mothers and their newborns during pregnancy. From April 3rd, 2020, to February 10th, 2023, data on 8,540 women and their newborns were collected, with active participation from 130 out of 686 (19%) German obstetric hospitals. The study was approved by the ethics committees of the coordinating center (UKSH Kiel, AZ: D 451/20) and each participating hospital. Information about CRONOS has been published on the German Society of Perinatal Medicine´s website, www.dgpm-online.org, and the German Clinical Trials Registry (DRKS00021208). About 2,000 women agreed to be contacted again for further follow-up.

The CRONOS-Kids study focuses on child health and will study some of the intrauterine-exposed children longitudinally. As an increased rate of placentitis with a concomitant increased risk of stillbirth and preterm delivery has been seen in infections with the Alpha and Delta variants, women with an SARS-CoV-2 infection between January 2021 and December 2021, initially recruited in the five participating university hospitals, will be contacted.

Recruiting for CRONOS-Kids On each of the five research sites, women initially participating in CRONOS will be invited via email, letter, or by phone to participate in the CRONOS-Kids study.

Unexposed children and their parents will be invited to participate via their local pediatricians.

All women will be able to book appointments at their respective hospitals via a dedicated website (http://cronos-kids.de). The management of patient contact will be conducted exclusively by non-examiners. Pseudonymization will be used.

Study instruments All children will undergo examination by personnel specifically trained for this purpose. In order to assess potential motor and cognitive deficiencies, the M-ABC-2 and the ASQ-3 will be utilised. Furthermore, social-emotional aspects will be addressed using a specific SE-test.

Questions of a general nature will address the subjects of pregnancy, birth, and social circumstances, with a view to identifying potential sources of bias with regard to developmental delays.

Potential bias To circumvent any potential bias in the study, responsibility for patient contact and examinations will be allocated to different members of the research team. Personnel conducting neurodevelopmental testing will adhere to the principles of blinding, ensuring that they remain unaware of the subjects' exposure status.

We expect a bias in the participation of highly educated and German-speaking families. This is likely to affect both the exposed and non-exposed groups.

Statistical analysis The Marburg University research team will manage data refinement. Analysis will control for potential confounders such as children´s sex, weeks of gestational age at birth, asphyxia at birth and social circumstances.

To be able to measure a mean effect in an unpaired t-test with an alpha level of 0.05 and a power of 0.8 (Cohen's d = 0.5), 64 subjects per group are required, i.e

ELIGIBILITY:
Inclusion Criteria:

* Toddlers (age 33 to 60 months), who were exposed (case) or not exposed (controll) with SARS-CoV-2 intrauterin.

Exclusion Criteria:

* No parental consent

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: In a pilot study intrauterine exposed toddlers are eligible for inclusion in the study if their mothers are registered in the CRONOS registry in the following five university hospitals: Marburg University Hospital, Jena University Hospital, Kiel University Hospital, Dresden University Hospital and Freiburg University Hospital.
  Controls, i.e. infants who have not been exposed to SARS-CoV-2, are eligible for enrolment if they live in the proximity of the recruiting hospitals.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Motoric skills | 36 to 60 months old children
  Motoric skills will be measured using the M-ABC-2 ("global rate"), as well as parental self reports in the ASQ-3 (areas: "gross motor" and "fine motor") with age-specific cut-off values.

SECONDARY OUTCOMES:
Communication | 36 to 60 months old children
  Communication will be measured using parental self reports in the ASQ-3 (area: "communication") with age-specific cut-off values.
Personal-Social development | 36 to 60 months old children
  Personal-social development will be measured using parental self reports in the ASQ-3 (area: "personal-social") and self reports in the social-emotional questionaire, both with age-specific cut-off values.

CONTACTS AND LOCATIONS:
Locations (1):
- Philipps University of Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No
Participants did not agree in data sharing.

REFERENCES:
- [Background] Pecks U, Mand N, Kolben T, Rudiger M, Oppelt P, Zollkau J, Dempfle A; The CRONOS registry. SARS-CoV-2 Infection During Pregnancy-An Analysis of Clinical Data From Germany and Austria From the CRONOS Registry. Dtsch Arztebl Int. 2022 Sep 5;119(35-36):588-594. doi: 10.3238/arztebl.m2022.0266. PMID 35794736
- See also: This website has been created with the express purpose of providing patients with information regarding the study. — https://cronos-kids.de